CLINICAL TRIAL: NCT00337714
Title: A Parallel, Randomized Multicenter Comparison of Triple Lumen Central Venous Catheters Impregnated With Silver Nanoparticles (AgTive®) Versus Conventional Catheters in Intensive Care Unit Patients
Brief Title: Comparison of Central Venous Catheters With Silver Nanoparticles Versus Conventional Catheters
Acronym: NanoAgCVC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: ISS, Dip.Tecnologie e Salute, Prof. Gianfranco Donelli (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 60% MURST no. 7020119-1
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2008-09

CONDITIONS: Central Venous Catheter Related Infections
Keywords: Central venous catheter,; bloodstream infections,; intensive care unit
MeSH Terms: conditions — Sepsis | interventions — colloidal silver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): in this arm conventional CVCs will be inserted
  Interventions: Procedure: CVC cannulation
- B (Active Comparator): group B will receive medicated silver nanoparticles CVC
  Interventions: Procedure: CVC impregnated with silver nanoparticles (AgTive®)

INTERVENTIONS:
Procedure: CVC impregnated with silver nanoparticles (AgTive®) — insertion of medicated silver nanoparticles CVC
  Arms: B
Procedure: CVC cannulation — placement of conventional trilumen CVCs
  Arms: A

SUMMARY:
Bloodstream infections are common in Intensive Care Units (ICUs). The need of a central venous line increases the risk of bacteremia and central venous catheter (CVC) related infections. The use of catheters coated and/or impregnated with different antimicrobial agents has been proposed to reduce the risk of such infections. However, results obtained so far did not reach enough clinical relevance to consider these medicated catheters as a valid alternative to the conventional ones.

The aim of this comparative randomized study is to assess the ability of recently developed silver ion-releasing central venous catheters in preventing associated infections in comparison with the conventional ones.

Experimental groups are defined as follows:

* Group A: patients treated with standard, triple lumen, non medicated catheters
* Group B: patients treated with triple lumen catheters impregnated with silver nanoparticles

DETAILED DESCRIPTION:
RATIONALE

Central venous catheter (CVC) infections are one of the major causes of infections acquired in intensive care unit (ICU) patients. About 25% of bloodstream infections recorded in ICUs are secondary to proven catheter-related infections and up to 80% of the so-called primary bacteraemia may be caused by catheters. Pittet et al. have estimated that nosocomial bloodstream infection, irrespective of its source, was associated with an overall 35% attributable mortality and a prolonged hospital stay of 32 days, including 8 days in the ICU. Prevention of catheter-related infections is a priority for infection control programs. Clear preventive measures include strict barrier precautions during insertion and careful aseptic techniques during subsequent manipulations of catheters. Other preventive measures, including the use of catheters specifically designed to inhibit microbial colonisation, such as antimicrobial-coated catheters, are not universally accepted or recommended for routine use, also due to their high cost. Previous trials have demonstrated a 50% risk reduction of infection rates when using antiseptic-coated catheters; however, their efficacy in reducing catheter related bloodstream infections is still unclear. A new generation of silver nanoparticle impregnated CVCs (Logicath AgTive®, Medex Medical INC., UK), has become recently available, but no clinical trial documenting their activity in preventing microbial colonization of catheters has been carried out so far. In this study, we want to assess the ability of this new generation catheters to prevent short-term (< 28 days) catheter-related infections in critically ill patients, in comparison with conventional untreated catheters.

STUDY POPULATION

All consecutively admitted critically ill patients needing central venous catheterization for more than 5 days.

TRIAL OBJECTIVE AND PURPOSE

The objective of this study is to test the ability of these new medicated catheters, to reduce the risk of Central Venous Catheter Related Infections (CVCRI) in ICU patients. CVCRI is defined as a positive culture from the catheter when hemoculture is concurrently positive for the same microbial strain for at least two consecutive times.

TRIAL DESIGN

Study Design

This is a randomized, open, controlled, parallel multicenter study involving 5 Italian ICUs and the supporting clinical microbiology laboratories under the supervision of Prof. Massimo Antonelli, for the clinical issues and Prof Gianfranco Donelli, for the microbiology issues. Statistical evaluation of the data will be under the responsibility of Dott. Andrea De Gaetano, belonging to the Biomatematic Laboratory of the Italian National Research Council (CNR-IASI).

Endpoints

The primary end-point is the difference in raw percentage occurrence of CVCRI (on a patient basis) between groups A and B.

The secondary end-point are the infection-free time and the probability of CVCRI as a function of multiple predictors.

METHODS

Randomization and blinding

An Internet-based randomization scheme, stratified by center, age and gender will be employed, indicating the allocated treatment at the moment of enrollment. The randomization procedure will require that when guide wire exchange is performed, a catheter from the same allocation group (medicated or not medicated) is used. The treatment will be open to the physician performing the procedure, and data collection will indicate group membership as A and B in random order. While the data manager will hold the key to the group/treatment associations, both the adjudication committee members (deciding on database record freezing) and the statisticians performing the analyses will be blinded to treatment allocation.

Insertion and maintenance of catheters

Recommendations will be provided to study centers to comply with maximal barrier precautions during insertion and repositioning of catheters, if indicated. A transparent, semipermeable dressing, will be provided to all the participating ICUs to be used after insertion, to allow daily inspection of the insertion site. Subsequent dressings will be carried out as clinically indicated, at 2 to 5 days intervals. Line tubing and three-way stopcocks will be changed on the basis of each unit's protocol at 1 to 3 days intervals, although changing these after each blood product transfusion and following the administration of lipid solutions will be required.

The catheter will be kept in place as long as required in the absence of complications. Catheters will be removed when no longer required, or because of malfunction, when suspicion of infection or otherwise unexplained bloodstream infection occurs; and in the presence of gross inflammation or pus at the catheter insertion site. In situ treatment of catheter infection will not be allowed.

Data recorded

The following information will be recorded upon inclusion: age, sex, date of hospital admission and to the intensive care unit; underlying disease and severity (McCabe class); admission category (medical, surgical, whether or not scheduled, or trauma), diagnosis and primary organ failure on ICU admission. The severity score SAPS II, organ dysfunction and SOFA score will also be recorded, as well as the presence of an active infection focus, ongoing antibiotic therapy, and presence of other intravascular devices. Patients will be followed up to 48 hours after catheter removal. Data recorded will include: a) Mechanical complication occurring during insertion (number of venipunctures, arterial puncture, hematoma, pneumothorax); b) presence of local signs suggesting infection (erythema at the catheter skin entry site, scored as 0: absence; 1+: <5mm; 2+: 5-10mm; 3+: >10mm; presence of induration or purulence); c) presence of a systemic inflammatory response syndrome or of symptoms characterizing severe sepsis; d) Presence of other documented infection ; e) other intravascular devices in place or inserted each day; f) dressing changes; g) Results of blood and catheter-tip cultures, and of other clinically significant microbiological samplings; h) antibiotics administered.

Microbiological data

Blood cultures will be obtained when temperature is > 38°2 or < 36°5C. Diagnostic samples of any other suspected infection foci will be taken as clinically indicated. Upon catheter removal, the intravascular catheter tip will be cultured using the semi quantitative culture described by Maki et al. (Maki DG, Weise CE, Sarafin HW. A semiquantitative culture method for identifying intravenous-catheter-related infection. N Engl J Med 1977;296:1305-1309). This technique involves rolling of the catheter distal tip on Agar plate and reading the high-density colonization on a semiquantitative culture (more than 15 colonies on each plate).

Inclusion Criteria

Patients will be eligible when insertion of a central venous catheter (CVC) at a new site (subclavian or internal jugular) has to be planned for therapy or monitoring of at least 3-day duration.

Exclusion Criteria Age below 18 years and all patients with a history of failed catheterization attempts or the need for catheterization at a site of previous surgery, skeletal deformity, or scarring.

Data analysis

A Clinical Evaluation (Adjudication) Committee composed of the two coordinating investigators (Prof. Massimo Antonelli and Prof. Gianfranco Donelli) and the statistician (Dr. Andrea De Gaetano) will assess, blindly with respect to the randomization group, the evaluability of catheters and the classification of all episodes of bloodstream infection and of catheters having a positive culture, according to the above definitions. Catheters will be excluded from the analysis when insertion fails. Catheters that have not been adequately followed-up until the time of removal (transfer to another unit or hospital) will be censored on the last day of follow-up in the ICU and classified by the Committee as infected or uninfected, using the data available up to the last day of follow-up and any bacteriological data subsequently received.

ASSESSMENT OF SAFETY

Adverse Events

Complications of the procedure will be classified according to a Complications Diagnosis Dictionary. Text comments will be added to the recordings as appropriate. Descriptive analysis of the complications as well as comparison of complication rates (overall and by family of most frequent complications) will be obtained.

STATISTICS

Sample Size and Power Computation

The catheter-related infection rate was estimated at 10% in the conventional catheter group. Assuming a 50% relative reduction (to 5%) in the silver impregnated CVC treated group, the number of patients needed (or equivalently the number of patients enrolled, assuming an attrition rate of 10%) for each treatment group in order to reach the desired statistical power is reported below, assuming a Type I error level of 0.05 and depending on the significance level and the number of tails of the statistical test.

Two-tailed tests will be considered throughout. A power of 80% will be considered sufficient. Therefore, 472 patients per group should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible when insertion of a central venous catheter (CVC) at a new site (subclavian or internal jugular) has to be planned for therapy or monitoring of at least 3-day duration.

Exclusion Criteria:

* Age below 18 years and all patients with a history of failed catheterization attempts or the need for catheterization at a site of previous surgery, skeletal deformity, or scarring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2006-07; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary end-point is the difference in raw percentage occurrence of central venous catheter related infections (CVCRI) (on a patient basis) between groups A and B. | period during the ICU stay

SECONDARY OUTCOMES:
The secondary end-point are the infection-free time and the probability of CVCRI as a function of multiple predictors. | period during the ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, Prof, Study Chair — Catholic University of the Sacred Heart
Locations (1):
- UCSC, Policlinico Universitario A. Gemelli, ICU, Rome, Rome, Italy

REFERENCES:
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT00337714